CLINICAL TRIAL: NCT05288595
Title: TCR Alpha/Beta and CD19-depleted Allogeneic Hematopoietic Cell Transplant for Malignant and Non-Malignant Disease
Brief Title: TCR Alpha/Beta and CD19-deplete Haplo-HSCT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Cancelled by Sponsor
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-2336.cc
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Patients; Hematologic Malignancy; Other Hematologic Condition
Keywords: Donor; granulocyte stimulating factor (GCSF); apheresis
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible Patients with a hematologic disease who could benefit from HCT with an eligible mismatched related or unrelated donor per donor selection criteria. Patient/recipient admitted of HCT/start of preparative regimen and stem cell infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Pediatric patients with malignant or non-malignant hematologic condition (Experimental): The infusion of the final TCRαβ/CD19 depleted product will be given through the recipient's central venous catheter and will be administered fresh, without cryopreservation whenever possible. If the product must be cryopreserved and then thawed, this will be done according to institutional standards.
  Interventions: Device: CliniMACS Plus Instrument

INTERVENTIONS:
Device: CliniMACS Plus Instrument — Miltenyi Biotec's CliniMACS Plus Instrument is to be used to TCRαβ CD19 deplete products utilized in this protocol. The CliniMACS Plus is an automated cell separation platform which is functionally closed, maintaining a sterile system for cell depletion and enrichment utilizing a magnetic separation column. Reagents and supplies are to be used for research only but are manufactured and tested under a quality system certified to ISO 13485. Should CD34 selection be required to augment stem cell dose, Miltenyi Biotec's CliniMACS® Plus CD34 Reagent System is FDA approved as a Humanitarian Use Device (HUD). The approved indication was the treatment of patients with acute myeloid leukemia (AML) undergoing myeloablative transplant from matched related allogeneic donors. The CliniMACS® Plus reagent system was approved to obtain an enriched CD34+ cell population for hematopoietic reconstitution without the need for GVHD prophylaxis.

SUMMARY:
This is an open label, interventional, non-randomized, phase II trial of TCR alpha/beta and CD19-depeleted allogeneic HCT in pediatric patients with hematologic disease.

DETAILED DESCRIPTION:
This is a single-site, open label, interventional, non-randomized, phase II trial of TCRαβ/CD19 deplete allogeneic HCT as donor source and sole GVHD prophylaxis in pediatric patients with either malignant or non-malignant hematologic disease who are eligable for allogeneic HCT, but lack a HLA-matched sibling donor.

ELIGIBILITY:
Inclusion Criteria:

1. Age 31 days to <30 years
2. Have a malignant or non-malignant hematologic disease, defined as disease resulting from abnormal function of a cell of the hematopoietic stem cell lineage, that could benefit from an allogeneic HCT. Examples include acute and chronic leukemias, myelodysplastic syndrome, lymphoma, severe acquired and congenital cytopenias/marrow failure, white blood cell abnormalities, red blood cell abnormalities, and platelet abnormalities.
3. Clinical remission for patients with acute leukemia (MDS/AML excluded) or lymphoma
4. Lack a healthy and willing HLA-identical related donor, with the exception of patients with FA who will be eligible with a willing HLA-identical related donor given the standard use of T-cell depletion in matched sibling donor HCT in FA
5. Have a related or an unrelated donor who meets the donor selection criteria, is healthy, willing, and able to receive GCSF with or without Plerixafor, and undergo apheresis through placement of catheters in the antecubital veins or a temporary central venous catheter
6. Able to give informed consent if ≥ 18 years, or with legal guardian capable of giving informed consent if < 18 years
7. Provision of signed and dated informed consent form

Exclusion Criteria:

1. Uncontrolled, active infection at time of HCT
2. HIV positivity
3. Cardiac ejection fraction <45%
4. Creatinine clearance <60 mL/min/1.72 mL
5. Pulmonary diffusion capacity (adjusted for hemoglobin), FEV1, or FVC <60% of predicted or an O2 saturation <94% on room air if unable to perform pulmonary function testing
6. Serum ALT >5x upper limit of normal or bilirubin >2
7. Performance score (Lansky or Karnofsky) <50
8. Pregnant or lactating females, as many medications necessary for a successful HCT are potentially harmful to unborn babies and infants.

Ages: 31 Days to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe (grade III-IV) acute graft-versus-host disease (GVHD) at day 100 after infusion of a TCRαβ+/CD19+ negative, peripheral blood stem cell (PBSC) product without additional GVHD prophylaxis. | 5 years
  Grade to be determined using Acute GVHD Staging Scale

SECONDARY OUTCOMES:
Number of patients with non-engraftment | 100 days
  Defined as the lack of donor-derived neutrophil engraftment
Number of patients with relapse | 1 year
  Interval from transplant to relapse/recurrence of disease
Number of treatment-related mortality (TRM) | 1 year
  Defined as death due to regimen-related toxicity or GVD.
Disease-free Survival (DFS) measured in days | 1 year
  Defined as the minimum time interval from transplant to relapse/recurrence of disease, death or last follow-up.
Overall Survival (OS) measured in days | 1 year
  Determined at 1 year post-HCT
Immune Reconstitution | 1 year
  Incidence of absolute CD4+ T-cell count >400 cells at 1 year post-HCT
Post-HCT infections | 100 days
  Incidence of bacterial, fungal, and viral infections at day +100

CONTACTS AND LOCATIONS:
Overall Officials: Alisa B Lee Sherick, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No